CLINICAL TRIAL: NCT06552000
Title: Phase 0 Trial of Pre-operative Tumor Treating Fields in Patients With Resectable Lung Cancer
Brief Title: Pre-operative Tumor Treating Fields in Patients With Resectable Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, John Waters, Assistant Professor, Cardiovascular & Thoracic Surgery, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC 07524; STU-2024-0624
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tumor Treatment Fields (Experimental): Duration: 2-4 week; target 18 hours/day (on average). Continuous between time of enrollment and date of surgery.
  Cycle Length: 2-4 weeks
  Interventions: Device: NovoTTF-200T System

INTERVENTIONS:
Device: NovoTTF-200T System — Exposure/Frequency: 150 kHz Route: Transdermal through patented microarray system to the hemithorax affected with cancer, 2-4 week duration, target 18 hours/day (on average)

SUMMARY:
The purpose of this study is to study the clinical and biologic effects of Tumor Treatment Fields (TTFields) in patients undergoing resection of stage I-IIIA Non-Small Cell Lung Cancer (NSCLC). TTField is a non-invasive treatment that uses low-intensity electrical fields to treat cancer. Resection is the medical term for surgically removing part or all of a tissue, structure, or organ.

DETAILED DESCRIPTION:
To study the clinical and biologic effects of Tumor Treatment Fields (TTFields) in patients undergoing resection of stage I-IIIA NSCLC.

Participants in this study will have a blood sample collected as well as vital signs along with a tumor tissue sample and tumor scan. Once it has been determined the participant can enroll into this study, he/she will come to the clinic for 5 scheduled visits over a period of 2 months .

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stage I-IIIA NSCLC planned for surgical resection.
2. Eastern Cooperative Oncology Group (ECOG) 0-2 performance status.
3. Willingness and ability to undergo planned correlative studies, including imaging tests.
4. Fresh biopsy diagnostic material obtained from standard of care procedure to perform baseline correlatives (10-15 slides)-if not available, enrollment will be considered on a case-by-case basis after discussion with and approval by the Lead Site PI or Lead Site Co-Principal Investigator.
5. Ability to understand and the willingness to sign a written informed consent.
6. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   * 6a. A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * • Has not undergone a hysterectomy or bilateral oophorectomy; or
   * • Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
7. Age ≥22 years at time of screening.

Exclusion Criteria:

1. Receipt of prior therapy for the current NSCLC.
2. Planned neoadjuvant therapy for the current NSCLC.
3. History of major allergic reactions attributed to adhesive or compounds in TTFields micro-array.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
5. Pregnant or nursing patients due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
6. Use of electronic devices or prosthetics - i.e., pacemakers, defibrillators, spinal infusion pumps. Specific scenarios can be discussed with the Lead Site PI or Lead Site Co-Principal Investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of TTF (Tumor-Treating Fields) on Fanconi anemia-related genes. | approximately 14-28 days
  Determine the effect of TTFields on expression of Fanconi anemia pathway-associated genes in NSCLC.

SECONDARY OUTCOMES:
Safety of administering TTFields | approximately 14-28 days
  Assess the safety of administering TTFields prior to standard of care lung cancer resection.
  Analyses will be performed for all subjects having initiated TTFields therapy. The study will use the CTCAE version 5.0 for reporting of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: John Waters, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No